CLINICAL TRIAL: NCT04933604
Title: Comparison of Laparoscopic Partial Nephrectomy Versus Laparoscopic Radical Nephrectomy in Patients With High-Complexity Renal Tumors: A Propensity Score Matched Analysis
Brief Title: LPN in Patients With High-complex Renal Tumors
Status: Completed | Type: Observational
Sponsor: Samsun Liv Hospital (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Mehmet Necmettin Mercimek, Principal Investigator, Samsun Liv Hospital
Other Study IDs: OMU KAEK 11.07.2019/538
Record Dates: First submitted 2021-05-31; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Renal Cancer; Renal Neoplasm; Renal Cell Carcinoma; Surgery; Oncology; Kidney Ischemia; Kidney Injury; Urologic Neoplasms; Urologic Cancer; Kidney Neoplasms
Keywords: Laparoscopy; nephrometry score; partial nephrectomy; propensity score matching; radical nephrectomy
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LPN group: 39 patients with high complexity renal tumors who underwent laparoscopic partial nephrectomy
  Interventions: Procedure: laparoscopic partial nephrectomy
- LRN group: 39 patients with high complexity renal tumors who underwent laparoscopic radical nephrectomy
  Interventions: Procedure: Laparoscopic radical nephrectomy

INTERVENTIONS:
Procedure: laparoscopic partial nephrectomy — Nephron sparing minimally invasive surgery
  Groups: LPN group
Procedure: Laparoscopic radical nephrectomy — Completely removal of kidney by using laparoscopic surgery
  Groups: LRN group

SUMMARY:
The study aims to investigate the rationale for LPN in patients with high-complexity renal tumors in terms of oncologic and functional outcomes.

DETAILED DESCRIPTION:
From November 2009 to October 2018, 399 patients underwent LPN and 307 patients to laparoscopic radical nephrectomy (LRN). 41 patients with RENAL score ≥ 10 enrolled in LPN and 265 patients to the LRN group. Propensity score matching (matched by age, gender, clinical tumor stage, tumor size, baseline renal function, comorbidities such as diabetes mellitus (DM), hypertension (HT), coronary artery disease (CAD), and final tumor pathology of RCC) was used to reduce selection bias. Functional and oncological outcomes were compared between the two groups. After propensity score analysis, 39 patients in the LRN group were matched with 39 in the LPN group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete data
* Patients with single renal tumor on the effected side
* Patients who approved the written consent form

Exclusion Criteria:

* Patients who not approved the written consent form
* Patients with incomplete data
* Patients with low or mild complexity renal tumors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From November 2009 to October 2018, 399 patients underwent LPN and 307 patients to laparoscopic radical nephrectomy (LRN). 41 patients with RENAL score ≥ 10 enrolled in LPN and 265 patients to the LRN group. Propensity score matching (matched by age, gender, clinical tumor stage, tumor size, baseline renal function, comorbidities such as diabetes mellitus (DM), hypertension (HT), coronary artery disease (CAD) and final tumor pathology of RCC) was used to reduce selection bias. Functional and oncological outcomes were compared between the two groups. After propensity score analysis, 39 patients in the LRN group were matched with 39 in the LPN group.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Operation time | at the end of the surgery
  time from onset to complete of surgery
Blood loss | at the end of the surgery
  amount of bleeding during surgery (mL)
warm ischemia time | at the and of the surgery
  The clamp time of the renal artery and vein which is required to complete tumor excision and renorrhaphy
Postoperative complication | up to 3 months postoperatively
  abnormal problmes that may be seen after surgery and require additional intervention, treatment or follow-up
functional outcomes | 1 year after the surgery
  serum creatinine level (mg /dL) and estimated glomerular filtration rate (CKD Epidemiology Collaboration (CKD-EPI) equation) (mL/min/1.73 m2)
surigcal margin status | postoperative follow-up, through study completion, an average of 1 year
  presence or absence of tumors at the surgical margin
CKD stage upgrading | postoperative follow-up, through study completion, an average of 1 year
  evaluation of preoperative and postoperative renal functions according to chronic kidney disease stages
Oncological outomes | postoperative follow-up, through study completion, an average of 1 year
  Presence or absence of local and/or distal tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Ender Ozden, Prof., Study Director — Ondokuz Mayıs Üniversitesi, Tıp Fakültesi, Üroloji Anabilim dalı; Saban Sarıkaya, Prof., Study Chair — Ondokuz Mayıs University, Faculty of Medicine, Department of Urology; Mehmet Mercimek, MD, FEBU, Principal Investigator — Liv Hospital Samsun, Department of Urology; Yakup Bostancı, Prof., Principal Investigator — Ondokuz Mayıs University, Faculty of Medicine, Department of Urology; Murat Gulsen, MD, Principal Investigator — Samsun Gazi State Hospital, Departmen of Urology, Samsun, Turkey
Locations (1):
- Ondokuz Mayıs University, Department of Urology, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kim SP, Campbell SC, Gill I, Lane BR, Van Poppel H, Smaldone MC, Volpe A, Kutikov A. Collaborative Review of Risk Benefit Trade-offs Between Partial and Radical Nephrectomy in the Management of Anatomically Complex Renal Masses. Eur Urol. 2017 Jul;72(1):64-75. doi: 10.1016/j.eururo.2016.11.038. Epub 2016 Dec 14. PMID 27988238
- [Result] Mir MC, Derweesh I, Porpiglia F, Zargar H, Mottrie A, Autorino R. Partial Nephrectomy Versus Radical Nephrectomy for Clinical T1b and T2 Renal Tumors: A Systematic Review and Meta-analysis of Comparative Studies. Eur Urol. 2017 Apr;71(4):606-617. doi: 10.1016/j.eururo.2016.08.060. Epub 2016 Sep 7. PMID 27614693
- [Result] Yang F, Zhou Q, Xing N. Comparison of survival and renal function between partial and radical laparoscopic nephrectomy for T1b renal cell carcinoma. J Cancer Res Clin Oncol. 2020 Jan;146(1):261-272. doi: 10.1007/s00432-019-03058-z. Epub 2019 Nov 1. PMID 31677114